CLINICAL TRIAL: NCT02359916
Title: Time Over Money? A Novel System to Influence Snack Machine Choices
Brief Title: Delays to Influence Snack Choice
Acronym: DISC
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Brad Appelhans, Associate Professor, Rush University Medical Center
Other Study IDs: 13012802
Record Dates: First submitted 2015-02-02; First posted 2015-02-10 (Estimated); Results first posted 2018-01-26 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Food Choice

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- A: Snacks sold under equal pricing, no delays
- B: Healthier snacks sold at 25% or $0.25 discount, no delays
  Interventions: Other: 25%/$0.25 discount on healthy snacks
- C: Less healthy snacks sold at equal pricing with delays
  Interventions: Other: Time delays on delivery of less healthy snacks
- D: Healthy snacks sold at 25% or $0.25 discount, plus delays on less healthy snacks
  Interventions: Other: Time delays on delivery of less healthy snacks; Other: 25%/$0.25 discount on healthy snacks
- E: Less healthy snacks sold at 25% or $0.25 higher price, no delays
  Interventions: Other: 25%/$0.25 tax on less healthy snacks
- F: Less healthy snacks sold at 25% or $0.25 higher price, plus delays
  Interventions: Other: Time delays on delivery of less healthy snacks; Other: 25%/$0.25 tax on less healthy snacks
- G: Snacks sold under equal pricing, no delays

INTERVENTIONS:
Other: Time delays on delivery of less healthy snacks
  Groups: C; D; F
Other: 25%/$0.25 discount on healthy snacks
  Groups: B; D
Other: 25%/$0.25 tax on less healthy snacks
  Groups: E; F

SUMMARY:
The pervasiveness of high-calorie, nutrient-poor snacks in the environment is believed to have contributed to the epidemic levels of obesity and cardiometabolic disease in the U.S. This project tests whether a novel snack vending machine system that uses brief time delays to reduce the immediacy of reward from unhealthy snacks will improve the healthfulness of snack choices. If successful, this project will identify a new environmental intervention that could contribute substantially to obesity and cardiometabolic disease prevention efforts in schools, worksites, and other settings.

DETAILED DESCRIPTION:
Environmental interventions that address the high availability of unhealthy snacks in the environment are needed to prevent a large projected increase in the incidence of obesity and cardiometabolic disease in the U.S. Prior studies from the investigators group and others suggests that the human preference for immediate gratification from food drives dietary overconsumption, but this knowledge has not yet translated to more effective dietary intervention strategies. This project tests whether a novel snack vending machine system that uses brief time delays to reduce the immediacy of reward from unhealthy snacks will improve the healthfulness of snack choices. This study uses an experimental design to compare brief time delays, two forms of 25% differential pricing, and time delays combined with both forms of 25% differential pricing on their ability to increase purchasing of healthy snacks. Test machines will be placed in existing, high-volume vending locations, and each of these five experimental conditions will run for roughly four weeks. Additionally, baseline purchasing under no intervention will be monitored for four weeks before and four weeks after the five experimental conditions. Specific Aim 2 compares the effects of these five interventions against baseline on the proportion of total vending sales from healthy snacks. Specific Aim 3 tests whether time delays or differential pricing harm overall vending machine sales in the test machines. This study not only tests a compelling theory about the effects of time delays and immediate reward on food choice, but evaluates the efficacy and feasibility of a novel intervention to improve the healthfulness of snack choices in worksites, schools, and other settings.

ELIGIBILITY:
Inclusion Criteria:

* Not applicable

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This is an environmental intervention. No subjects will be recruited or enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 32662 (Actual)
Dates: Start 2015-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley M Appelhans, PhD, Principal Investigator — Associate Professor
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Appelhans BM, French SA, Olinger T, Bogucki M, Janssen I, Avery-Mamer EF, Powell LM. Leveraging delay discounting for health: Can time delays influence food choice? Appetite. 2018 Jul 1;126:16-25. doi: 10.1016/j.appet.2018.03.010. Epub 2018 Mar 15. PMID 29551401

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Vends
Groups:
- Baseline 1: Snacks sold under equal pricing, no delays. Baseline 1 was always the first condition at all vending sites.
- Discount Only: Healthier snacks sold at 25% or $0.25 discount, no delays
  25%/$0.25 discount on healthy snacks
- Delay Only: Less healthy snacks sold at equal pricing with delays
  25-second time delays on delivery of less healthy snacks
- Delay + Discount: Healthy snacks sold at 25% or $0.25 discount, plus delays on less healthy snacks
  25-second time delays on delivery of less healthy snacks
  25%/$0.25 discount on healthy snacks
- Tax Only: Less healthy snacks sold at 25% or $0.25 higher price, no delays
  25%/$0.25 tax on less healthy snacks
- Delay + Tax: Less healthy snacks sold at 25% or $0.25 higher price, plus delays
  Time delays on delivery of less healthy snacks
  25%/$0.25 tax on less healthy snacks
- Baseline 2: Snacks sold under equal pricing, no delays. Baseline 2 was always the last condition at all vending sites.
Period: Overall Study
Arm/Group | Baseline 1 | Discount Only | Delay Only | Delay + Discount | Tax Only | Delay + Tax | Baseline 2
Started (The unit of analysis for this study was vending machine sales ("vends").) | NA; 5481 Vends (The number of unique individuals in this study is unknown) | NA; 5784 Vends (The number of unique individuals in this study is unknown) | NA; 7473 Vends (The number of unique individuals in this study is unknown) | NA; 1996 Vends (The number of unique individuals in this study is unknown) | NA; 2846 Vends (The number of unique individuals in this study is unknown) | NA; 3438 Vends (The number of unique individuals in this study is unknown) | NA; 5644 Vends (The number of unique individuals in this study is unknown)
Completed | NA; 5481 Vends (The number of unique individuals in this study is unknown) | NA; 5784 Vends (The number of unique individuals in this study is unknown) | NA; 7473 Vends (The number of unique individuals in this study is unknown) | NA; 1996 Vends (The number of unique individuals in this study is unknown) | NA; 2846 Vends (The number of unique individuals in this study is unknown) | NA; 3438 Vends (The number of unique individuals in this study is unknown) | NA; 5644 Vends (The number of unique individuals in this study is unknown)
Not Completed | NA; 0 Vends | NA; 0 Vends | NA; 0 Vends | NA; 0 Vends | NA; 0 Vends | NA; 0 Vends | NA; 0 Vends

BASELINE CHARACTERISTICS:
Population: The unit of analysis for this study were vending machine sales ("vends"). No data was collected from individual participants. The number of unique individuals in this study is unknown.
Groups:
- Total: Total of all reporting groups
Arm/Group | Baseline 1 | Discount Only | Delay Only | Delay + Discount | Tax Only | Delay + Tax | Baseline 2 | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Customized — Age was not collected in this study
Sex/Gender, Customized — Sex/Gender was not collected in this study
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Healthy Snacks Purchased
Description: For each experimental condition, we will calculate the proportion of healthy vs unhealthy snacks sold over 4 weeks.
Time Frame: 28 weeks per vending location
Population: In this table, each vend is treated as an analyzed participant. No data were collected from individual human subjects. Analyses included all available data on healthy and regular snack vends. Data from Baseline 1 and Baseline 2 were combined into a single arm/group ("Baseline") in statistical analyses.
Measure: Number; unit: proportion of vends from healthy snacks
Units Other Than Participants: Vends
Groups:
- Baseline: Snacks sold under equal pricing, no delays. Data from Baseline 1 and 2 were combined in this analysis.
Arm/Group | Baseline | Discount Only | Delay Only | Delay + Discount | Tax Only | Delay + Tax
Number analyzed (Participants) | NA | NA | NA | NA | NA | NA
Number analyzed (Vends) | 11125 | 5784 | 7473 | 1996 | 2846 | 3438
proportion of vends from healthy snacks | .403 | .431 | .429 | .465 | .542 | .501

2. Secondary Outcome: Total Daily Vending Revenue in US$/Day
Description: Total vending machine revenue under each condition
Time Frame: Number of days per condition were as follows - Baseline: 119 days, Discount only: 59 days, Delay only: 68 days, Delay + Discount: 49 days, Tax only: 73 days, Delay + Tax: 60 days
Population: The unit of analysis is vending revenue per day ($/day). Data from Baseline 1 and Baseline 2 were combined into a single arm/group ("Baseline") in this analysis.
Measure: Mean (Standard Deviation); unit: $/day
Units Other Than Participants: Days
Groups:
- Baseline: Snacks sold under equal pricing, no delays
Arm/Group | Baseline | Discount Only | Delay Only | Delay + Discount | Tax Only | Delay + Tax
Number analyzed (Participants) | NA | NA | NA | NA | NA | NA
Number analyzed (Days) | 119 | 59 | 68 | 49 | 73 | 60
$/day | 45.4 (31.6) | 42.1 (33.3) | 44.6 (27.7) | 35.9 (21.0) | 46.4 (35.6) | 51.9 (66.5)

ADVERSE EVENTS:
Description: Adverse events were not collected in this study.
Arm/Group | Baseline | Discount Only | Delay Only | Delay + Discount | Tax Only | Delay + Tax
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No